CLINICAL TRIAL: NCT01435070
Title: A Correlation of Functional Outcome Measures of Fractures of the Distal Radius Following Operative Management
Brief Title: Functional Outcome Following Fracture of the Distal Radius
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Warwick (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other); DePuy International (Industry)
Responsible Party: Principal Investigator, Caroline Plant, Mrs Caroline Plant, University of Warwick
Other Study IDs: IIS2010025
Record Dates: First submitted 2011-08-30; First posted 2011-09-15 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Distal Radius Fractures
Keywords: Colles' fracture; Radius fracture; grip strength; pinch strength; range of movement; PRWE; DASH; EQ-5D; Kirschner wire; Volar locking plate
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture; Radius Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Bone Plates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Distal radius fracture: Patients aged 18 years and older with a fracture of the distal radius, within 3 cm of the radiocarpal joint
  Interventions: Procedure: Kirschner wire fixation; Procedure: Volar Locking Plate fixation

INTERVENTIONS:
Procedure: Kirschner wire fixation — The wires are passed through the skin over the dorsal aspect of the distal radius and into the bone in order to hold the fracture in the correct (anatomical) position. The size and number of wires, the insertion technique and the configuration of wires will be left entirely to the discretion of the surgeon.
  A plaster cast will be applied at the end of the procedure to supplement the wire fixation as per standard surgical practice. This cast holds the wrist still and is left on until the wires are removed at the follow-up appointment.
  Other Names: K-wire fixation
Procedure: Volar Locking Plate fixation — The locking-plate is applied through an incision over the volar (palm) aspect of the wrist. The surgical approach, the type of plate and the number and configuration of screws will be left to the discretion of the surgeon. The screws in the distal portion of the bone will be fixed-angle, i.e. screwed into the plate, but this is standard technique for use of these plates. The type of proximal screw will be left to the discretion of the surgeon; these may be locking or non-locking screws. The use of a cast will left to the discretion of the surgeon.
  Other Names: open reduction and internal fixation; plate and screw fixation

SUMMARY:
Patients attending the University Hospital Coventry UK with a broken wrist requiring an operation, will be invited to enter the study. At the first visit, they will have an xray of the wrist and will be asked to complete a number of questionnaires. The questions are to determine if they normally have pain in the wrist and how well they can perform their daily activities. The patient will then have an operation, and the fracture in the wrist will be held in the correct position with either a metal plate and screws or wires.

At 6 weeks following the operation the patient will be reassessed and an xray will be taken. At 3 months, 6 months and 12 months after the operation patients will perform tests to assess the strength of their grip, pinch and movement of their wrist. In addition they will complete the the same questionnaires from their first visit. At the 12 month visit patients will have another xray.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a dorsally displaced fracture of the distal radius, which is defined as a fracture within 3cm of the radio-carpal joint
* The treating Consultant surgeon believes that they would benefit from operative fixation of the fracture
* Aged over 18years (either sex) and able to give informed consent

Exclusion Criteria:

* The fracture extends more than 3 cm from the radio-carpal joint
* The fracture open with a Gustillo grading greater than 1
* There are contra-indications to general anaesthetic
* There is evidence that the patient would be unable to adhere to trial procedures or complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to University Hospital Coventry with an acute fracture of the distal radius requiring operative management
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 1 year post-operatively
  Maximum grip strength applied to a hand-held dynamometer, measured in kilograms

SECONDARY OUTCOMES:
Pinch strength | 1 year post-operatively
  The force in kilograms of the pinch between the thumb pad and the radial aspect of the middle phalanx of the index finger when applied to a pinch gauge.
Wrist arc motion | 1 year post-operatively
  The range of motion in flexion-extension, radioulnar deviation and supination-pronation of the wrist and forearm.
Patient rated wrist evaluation (PRWE) | 1 year post-operatively
  The PRWE score is a validated self-reported questionnaire. It consists of 15 items specifically related to the function of the wrist.
Disabilities of Arm, Shoulder and Hand Score (DASH) | 1 year post-operatively
  The DASH outcome measure is a 30-item, self-report questionnaire designed to provide a more general measure of physical function and symptoms in people with musculoskeletal disorders of the upper limb
EQ-5D | 1 year post-operatively
  A validated, generalised, quality of life questionnaire consisting of 5 domains related to daily activities with a 3-level answer possibility. The combination of answers leads to the QoL score.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Costa, FRCS, PhD, Study Chair — Warwick Orthopaedics; Juul Achten, PhD, Study Director — Warwick Orthopaedics; Caroline E Plant, BSc, MBChB, Principal Investigator — Warwick Orthopaedics
Locations (1):
- Warwick Medical School, Coventry, Warwickshire, United Kingdom